CLINICAL TRIAL: NCT01286623
Title: Study Title: The Pharmacology/Aging Clinic: Clinical Routine Monitoring of HIV-infected Patients Over 50 Year of Age.
Brief Title: The Pharmacology/Aging Clinic
Acronym: SSAT041
Status: Completed | Type: Observational
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SSAT 041
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The treatment of HIV and the tests performed for HIV care have changed over the last 20 years. However, improvement of management of HIV-infected subjects is still warranted, especially as the HIV-infected population is aging. Therefore, this study will involve the collection and analysis of clinical information obtained from subjects who are over 50 years of age. For example, patients' risk of heart disease will be measured and monitored by looking at blood tests and clinical data (such as blood pressure). This will allow researchers to understand if the current way of assessing the risk of future heart disease is the best one available for HIV-infected individuals. No genetic research will be done.

DETAILED DESCRIPTION:
Patients will be asked to read the information contained in this leaflet. No extra visits will occur; all samples will be collected at their routine visits to the pharmacology clinic. All blood samples and results will be managed by the routine clinical laboratory at Chelsea and Westminster Hospital, with the exception of the assessment of the hsCRP. The latter is a marker of inflammation that is measured to be able to add more information when cardiovascular risk is assessed. The blood sample for this test is sent to a laboratory in London called The Doctors Laboratory (TDL). All shipped samples are anonymous and patient names will not be disclosed outside the Hospital.

The clinical visits will be scheduled approximately once within one year. However, extra visits may be clinically necessary if a clinical condition requires proper follow-up. Furthermore, clinical details will be marked to show patients have agreed to their use for this research study.

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form
2. HIV-infected patients attending the Pharmacology/Aging Clinic (HIV/GUM Directorate, Chelsea and Westminster Hospital NHS Foundation Trust)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected patients over 50 years of age
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2013-06-06 (Actual); Study Completion 2013-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Boffito, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's Centre, London, United Kingdom